

File type: Subject Informed Consent Form

**Official title:** Evaluating the efficacy of a text messaging-based shisha smoking cessation intervention for young adults in Hong Kong: a randomised controlled pilot trial

NCT number: NCT ID not yet assigned

**Document Date:** 25<sup>th</sup> August 2024



## **Subject Informed Consent Form**

Title of study: Evaluating the efficacy of a text messaging-based shisha smoking cessation intervention for young adults in Hong Kong: A pilot randomised controlled trial.

| Subject identification number: SSCI-E – | | | | |
|---|---|---|---|---|
| 1. | I confirm that I have read and understood | I the information sheet for the ab | nove | П |
| study and have had the opportunity to ask questions. | | | 0,0 | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw | | | |
| | at any time, without giving any reason. | | | |
| 3. | . I understand that sections of any of my research notes may be looked at by the | | | |
| | responsible regulatory authorities where it is relevant to my taking part in the | | | |
| | research I give permission for these parties to have access to my records. | | | |
| 4. | I understand and permit the data collected in this study to be used for publication | | | |
| _ | in academic journal without me being identified individually. | | | |
| 5. | 5. I agree to take part in the above study. | | | Ц |
| Resear | cher's Name: | Signature: | _ Date: | |
| Subjec | t's name: | Signature: | _ Date: | |
| Copies to: subject □ Researcher's file □ | | | | |

last updated: 25 Aug 2024